CLINICAL TRIAL: NCT06565364
Title: Immunogenicity and Thrombotic Potential of Circulating Protamine-heparin Complexes in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Caroline Holaubek, MD, Medical Doctor, Research Fellow, Medical University of Vienna
Other Study IDs: EK Nr: 1895/2014
Record Dates: First submitted 2024-08-07; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Thrombocytopenia; Antibodies Drug Specific
Keywords: Thrombin generation; Protamine
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: "ZYMUTEST™ HIA" immunoglobulin g ELISA (enzyme-linked immunosorbent assay ) — The enzyme-linked immunosorbent assay is an in vitro test done in the laboratory to detect specific antibodies against heparin/platelet factor-4 and protamine/heparin complexes.

SUMMARY:
The primary aim of this study was to describe the prevalence and time course of the occurrence of protamine/heparin antibodies in patients undergoing cardiac surgery on cardiopulmonary bypass.

The second aim was to identify triggers of immunization.

The third aim of this study was to evaluate a potential clinical impact of protamine/heparin antibodies and their platelet-activating properties leading to thromboembolism and other adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* cardiac surgery on cardiopulmonary bypass

Exclusion Criteria:

* cardiac surgery without cardiopulmonary bypass
* age < 18 years
* no written consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 160 patients were included to the study with written informed consent. 4 patients did not undergo the planned surgical procedure due to medical reasons and therefore had to be excluded subsequently.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
prevalence of protamine/heparin antibodies | preoperatively until postoperative day 10

SECONDARY OUTCOMES:
Potential triggers | preoperatively
  The presence of the following conditions was evaluated preoperatively:
  * repeated surgery on cardiopulmonary bypass (CPB)
  * bleeding disorders
  * age in years
  * height in meters
  * weight in kilograms
  * weight and height will be combined to report the body-mass-index in kg/m^2
  * previous thromboembolic event
  * diabetes mellitus with/without insulin treatment
  * cardiac function and valve diseases
  * preoperative presence of peripheral artery disease
  * preoperative presence of renal diseases
  * fish allergy
  * men after vasectomy
Clinical impact | until postoperative day 10
  Information about the following events were collected until day 10 or discharge of the patients:
  * cardiovascular events: thrombosis, tachycardic atrial fibrillation, cardiopulmonary resuscitation
  * delay in platelet count recovery
  * difference in severity of thrombocytopenia (platelet count in 10^9/l)
  * cerebrovascular events: stroke, seizure
  * kidney function: creatinine in mg/dl, urea in mg/dl, need for renal replacement therapy
  * inflammation parameters: white blood count in 10^9/l, C-reactive protein in mg/dl

OTHER OUTCOMES:
Thrombin generation | preoperatively until postoperative day 6
  measurement of thrombin generation in a reduced number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Steinlechner, MD, Principal Investigator — Department of Anaesthesia, Intensive Care Medicine and Pain Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Due to an ongoing Doctor of Philosophy (PhD) Thesis the dataset is not available at the moment